CLINICAL TRIAL: NCT00440635
Title: International Single-Arm Protocol to Provide Expanded Access to Bortezomib for Patients With Multiple Myeloma Who Have Received at Least 2 Previous Lines of Therapy and Are Refractory to or Have Relapsed After Their Last Therapy for Multiple Myeloma
Brief Title: Expanded Access Protocol (EAP) to Provide Bortezomib to Patients With Multiple Myeloma Who Have Received at Least 2 Previous Lines of Therapy and Are Refractory to or Have Relapsed After Their Last Therapy for Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag International NV (Industry)
Other Study IDs: CR002185
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; bortezomib, Hematology
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Drug: Bortezomib, tradename Velcade

SUMMARY:
The purpose of this study is to provide bortezomib to patients with multiple myeloma who have received at least 2 previous lines of therapy and are refractory or have relapse after their last treatment. Additional objectives of this study are assess the safety and tolerability of bortezomib and follow the levels of paraprotein in patients receiving bortezomib as a way to followup disease burden

DETAILED DESCRIPTION:
Multiple myeloma is uniformly fatal. Responses achieved after multiple lines of therapy are normally of short duration. Therefore, all patients with multiple myeloma will eventually relapse, having become refractory to therapy and subsequently will die of their cancer. The rationale of this study is that bortezomib as a novel agent may allow additional periods of response due to its different mechanisms of action. This is an open-label, single-arm, multicenter, non-comparative study to provide expanded access to bortezomib to patients with multiple myeloma that have received at least two previous lines of therapy and are refractory to or have relapsed after their last treatment. Patients will receive treatment with bortezomib 1.3 mg/m2 on day 1, 4, 8 and 11 of a 3-week cycle. No treatment will be administered on the last 10 days of each cycle. Treatment may be repeated for up to 8 cycles with possible extension if patient is still responding at the end of the 8 cycle period. Bortezomib 1.3 mg/m2 will be administered as an IV bolus

ELIGIBILITY:
Inclusion Criteria:

* Patients with previous diagnosis of multiple myeloma based on standard criteria
* patient has received at least 2 previous lines of therapy for multiple myeloma and, currently requires therapy because of relapsed or progressive disease
* If female, the patient is either postmenopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) from Screening through the Final Visit
* If male, the patient agrees to use an acceptable barrier method for contraception from Screening through the Final Visit
* patient has a Karnofsky performance status >= 60
* patient meets defined pretreatment laboratory criteria

Exclusion Criteria:

* If patient received bortezomib in a previous clinical trial, the patient's best response to bortezomib was progressive disease
* Patient received nitrosoureas within 6 weeks or any other chemotherapy within 3 weeks before enrollment, corticosteroids (>10 mg/day prednisone or equivalent) within 3 weeks before enrollment, immunotherapy or antibody therapy within 4 weeks before enrollment
* Patient has peripheral neuropathy of Grade 2 or greater intensity, as defined by the NCI CTC
* Patient had a myocardial infarction within 6 months of enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Patient has cardiac amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2004-01; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV

REFERENCES:
- [Derived] Quach H, Horvath N, Cannell P, Mikhael JR, Butcher BE, Prince HM. Safety and efficacy results from an international expanded access programme to bortezomib for patients with relapsed and/or refractory multiple myeloma: a subset analysis of the Australian and New Zealand data of 111 patients. Intern Med J. 2009 May;39(5):290-5. doi: 10.1111/j.1445-5994.2008.01738.x. Epub 2008 Jun 28. PMID 19371392